CLINICAL TRIAL: NCT01952002
Title: CLINICAL SAFETY FOR THE INSPIRATORY MUSCLE TRAINING IN CARDIOPULMONARY REHABILITATION PROGRAM
Brief Title: Clinical Safety for the Inspiratory Muscle Training
Status: Completed | Type: Observational
Sponsor: Clínica de Medicina do Exercício (Other)
Responsible Party: Sponsor
Other Study IDs: 0166.0.000.399-11; 304328/2011-1 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Heart Diseases; Lung Disease
Keywords: Blood Pressure; heart rate; electrocardiogram; Cardiac arrhythmias; respiratory exercise
MeSH Terms: conditions — Heart Diseases; Lung Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IMT - Inspiratory Muscle Training: 21 (16 males/5 femalesen) with a mean age of 73 ± 7.4 years were studied. Among the 21 study participants, the most prevalent clinical condition was coronary artery disease (11 cases); four individuals showing a diagnosis of chronic obstructive pulmonary disease and/or asthma, two presented congestive heart failure and the last four had other diseases
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Each session The session itself consisted of the following: two sets of 15 breathe cycles without removing the breathing promoter from the mouth and with the aid of a nose clip and 1-minute interval between sets. For training, we used the breathing promoters Power Breathe® Plus Light and Medium Resistance, possessing 10 levels of load gradation ranging from 17 to 186 cm H2O, which were adjusted for each patient and allowed for the individualized prescription of IMT

SUMMARY:
The aim of this study is evaluate the clinical, hemodynamic and electrocardiographic responses during an inspiratory muscle training session during a single cardiopulmonary rehabilitation session program. An electrocardiogram will be continuously recorded and the heart rate (HR) and blood pressure (BP) will be evaluated before, during and immediately after a single inspiratory muscle training (IMT) session, consisting of two series of 15 cycles, with one-minute intervals between sets and an initial load of at least 30% of the initial maximal inspiratory pressure (MIP).

ELIGIBILITY:
Inclusion Criteria:

* Patients regularly attending a supervised exercise program
* Patients were already performing the IMT in their usual supervisioned exercise sessions

Exclusion Criteria:

* cognitive impairment

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients regularly attending a supervised exercise program
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
abnormal clinical responses | One day
  During an IMT session, with two sets of 15 cycles at 30% of the load observed in MIP, there were no significant clinical or hemodynamic changes in patients regularly attending a supervised exercise program. In contrast, there are relatively frequent inductions of cardiac arrhythmias, mostly of low complexity, and more rarely, fleeting changes in ventricular repolarization during an IMT session.

SECONDARY OUTCOMES:
hemodynamic (blood pressure and heart rate) responses | one day
electrocardiographic pattern changes | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimex - Clínica de Medicina do Exercício, Rio de Janeiro, Rio de Janeiro, Brazil